CLINICAL TRIAL: NCT04149730
Title: Adrenaline During Resuscitation From Pulseless Electrical Activity
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/785
Record Dates: First submitted 2019-10-18; First posted 2019-11-04 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Heart Arrest
Keywords: Epinephrine; Pulseless electrical activity
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary PEA.: Patients at St. Olavs hospital who suffer cardiac arrest and pulseless electrical activity (PEA) as primary rhythm during 2018-2021. 120 episodes from St. Olavs hospital were collected previously (2010-2013). In addition 200 cases will be available from the hospital of The University of Pennsylvania, Philadelphia, USA.

SUMMARY:
This is a prospective observational study at St. Olavs hospital in Norway. Data are gathered from defibrillators that have been in use during resuscitation from cardiac arrest. Aim is to investigate the changes in electrocardiograms (ECG) during resuscitation from pulseless electrical activity (PEA), which is a type of cardiac arrest. ECG changes may be useful as a prognostic marker during resuscitation from PEA. In addition the researchers will describe the effect of adrenaline and chest compressions on clinical state transitions during resuscitation from pulseless electrical activity. Clinical state transitions are changes between different types of cardiac arrest. This study is expected to increase our understanding of the dynamics during treatment of cardiac arrest.

ELIGIBILITY:
Inclusion Criteria: Cardiac arrest among hospitalized patients presenting with PEA as the primary rhythm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of patients suffering cardiac arrest while being hospitalized at St. Olavs hospital.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
QRS frequency | Every 3 minutes from start till end of cardiopulmonary resuscitation
  Measurement of RR intervals in milliseconds.
QRS width | Every 3 minutes from start till end of cardiopulmonary resuscitation
  Measurement of the width of QRS complexes in milliseconds
Changes of clinical states | Every 3 minutes from start till end of cardiopulmonary resuscitation
  changes of clinical states (for example from Pulseless electrical activity to Ventricular fibrillation) during treatment of cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Skogvoll, md prof, Study Director — St. Olavs Hospital
Locations (2):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No